CLINICAL TRIAL: NCT02082574
Title: Prevalence of Cerebral Small Vessels Disease (CSVD) Among Patients Infected With HIV-1
Brief Title: Prevalence of Cerebral Small Vessel Disease in HIV Infected Patients
Acronym: MICROBREAK1
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2013-6
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-07

CONDITIONS: HIV Seropositivity
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients: HIV infected for more than 5 years, aged over 50, treated with ARV
- control: non HIV (matched for age and gender)

SUMMARY:
Cerebral small vessel disease (CSVD) is a major cause of cognitive impairment and disability in the general population, secondary to the accumulation of asymptomatic elementary lesions. CSVD is directly correlated with age and cardiovascular risk factors and therefore would be challenging in term of public health care in the future. While HIV patients share the same cardiovascular risk factors and they are often diagnosed with cognitive impairment and frailty, CSVD has not been yet described in this population.

The global aim is to compare the prevalence of CSVD in a well controlled HIV+ population compared to HIV- controls matched with age and sex.

500 HIV+ patients and 250 age- and sex- matched controls will undergo a screening of the CSVD with a 10 minutes MRI (FLAIR and T2*).

Prevalence of the CSVD will be compared between HIV+ patients and controls. General and HIV-specific parameters from their electronic medical records will be compared between HIV+/CSVD+ and HIV+/CSVD- patients.

We are expecting to prove that CSVD is more frequent in HIV+ population.

ELIGIBILITY:
Inclusion Criteria:

* age over 50
* chronic HIV seropositive patient infected for at least 5 years
* treated with any antiretroviral (ARV) therapy
* plasmatic HIV viral load <40 copies/ml for at least one year with one authorized blip < 1000 copies/ml per year

Exclusion Criteria:

* co-infection with hepatitis C virus (HCV)
* uncontrolled high blood pressure (WHO criteria)
* Personal history of cerebral infarction or cerebral ischemia
* Personal history of neurological complication of the HIV-infection
* Use of illegal drugs (except cannabis or poppers)
* Glomerular filtration rate < 15 mL/mn
* Complicated diabetes mellitus (glomerular filtration rate < 60ml/mn and/or proteinuria> 300 mg and/or retinopathy)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients over 50 years old, infected for at least 5 years, treated with antiretroviral (ARV) therapy
Sampling Method: Non-Probability Sample
Enrollment: 655 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Cerebral small vessel disease | baseline
  Cerebral small vessel disease detected with MRI

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MOULIGNIER, Dr, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France